CLINICAL TRIAL: NCT00349232
Title: Prevalence of Overweight and Obesity in Children Attending Special Primary Education and the Effect of a Lifestyle Intervention.
Brief Title: Lifestyle Intervention in Obese Children Attending Special Primary Education.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College of Antwerp (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HA-KINE-2006-001
Record Dates: First submitted 2006-07-04; First posted 2006-07-06 (Estimated); Last update posted 2006-07-10 (Estimated); Status verified 2006-07

CONDITIONS: Overweight; Obesity
Keywords: childhood obesity; lifestyle intervention; school health program; special primary education
MeSH Terms: conditions — Overweight; Obesity; Pediatric Obesity | interventions — Diet; Exercise

INTERVENTIONS:
Behavioral: lifestyle intervention (diet and physical activity)

SUMMARY:
The purpose of this study is to assess the prevalence of overweight and obesity in children attending special primary education and to evaluate the effects of a multidisciplinary school-based lifestyle intervention.

DETAILED DESCRIPTION:
Lifestyle changes related to high-fat diets and low levels of physical activity have resulted in a rising prevalence of overweight and obesity in children and adolescents. Ten per cent of the world's school-aged children are estimated to have excess body fat. Overweight and obesity during childhood and adolescence tend to continue into adulthood, increasing the likelihood of a range of impaired health conditions including cardiovascular diseases, diabetes and some cancers. School-based interventions have been proposed to prevent or treat obesity and have been described as a promising approach to reducing obesity among youth. First the extent and the characteristics of the problem have to be assessed for different types of education.

Comparison(s): the prevalence of overweight and obesity in special primary education will be compared to the prevalence in regular primary education. In special primary education, obese and overweight children will be randomised into a experimentel group (6 months of lifestyle intervention including diet and physical activity) and a control group (6 months normal treatment, if any, e.g. exercises for motor skills).

ELIGIBILITY:
Inclusion Criteria:

* children attending special and regular primary education

Exclusion Criteria:

* endocrine conditions affecting bodyweight (e.g. thyroid disease, diabetes)
* mental or physical disabilities that make it impossible to participate in sports activities

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100
Dates: Start 2006-07; Study Completion 2007-07

PRIMARY OUTCOMES:
Bodyweight after 3 and 6 months
Bodycomposition after 3 and 6 months
Bodyfat distribution after 3 and 6 months

SECONDARY OUTCOMES:
Eating behavior after 3 and 6 months
Physical activity after 3 and 6 months
Quality of life after 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Truijen, PhD, Study Chair — University College of Antwerp; Luc Van Gaal, MD, PhD, Principal Investigator — Universiteit Antwerpen; Dirk Vissers, Study Director — University College of Antwerp
Locations (1):
- MPI Zonnebos, Antwerp, Antwerp, Belgium

REFERENCES:
- [Background] Lobstein T, Baur L, Uauy R; IASO International Obesity TaskForce. Obesity in children and young people: a crisis in public health. Obes Rev. 2004 May;5 Suppl 1:4-104. doi: 10.1111/j.1467-789X.2004.00133.x. No abstract available. PMID 15096099
- [Background] Hulens M, Beunen G, Claessens AL, Lefevre J, Thomis M, Philippaerts R, Borms J, Vrijens J, Lysens R, Vansant G. Trends in BMI among Belgian children, adolescents and adults from 1969 to 1996. Int J Obes Relat Metab Disord. 2001 Mar;25(3):395-9. doi: 10.1038/sj.ijo.0801513. PMID 11319638
- [Background] Must A, Strauss RS. Risks and consequences of childhood and adolescent obesity. Int J Obes Relat Metab Disord. 1999 Mar;23 Suppl 2:S2-11. doi: 10.1038/sj.ijo.0800852. PMID 10340798
- [Background] Goran MI. Metabolic precursors and effects of obesity in children: a decade of progress, 1990-1999. Am J Clin Nutr. 2001 Feb;73(2):158-71. doi: 10.1093/ajcn/73.2.158. PMID 11157310
- [Background] Van Gaal LF, Wauters MA, De Leeuw IH. The beneficial effects of modest weight loss on cardiovascular risk factors. Int J Obes Relat Metab Disord. 1997 Mar;21 Suppl 1:S5-9. PMID 9130034
- [Background] Gortmaker SL, Peterson K, Wiecha J, Sobol AM, Dixit S, Fox MK, Laird N. Reducing obesity via a school-based interdisciplinary intervention among youth: Planet Health. Arch Pediatr Adolesc Med. 1999 Apr;153(4):409-18. doi: 10.1001/archpedi.153.4.409. PMID 10201726
- [Background] Muller MJ, Danielzik S, Pust S. School- and family-based interventions to prevent overweight in children. Proc Nutr Soc. 2005 May;64(2):249-54. doi: 10.1079/pns2005424. PMID 15960869